CLINICAL TRIAL: NCT04287946
Title: Endovascular Ablation of the Greater Splanchnic Nerve in Subjects Having Heart Failure With Preserved Ejection Fraction - First In-human Feasibility Study
Brief Title: Endovascular GSN Ablation in Subjects With HFpEF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Axon Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08938
Record Dates: First submitted 2020-02-19; First posted 2020-02-27 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure; Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Ablation (Experimental)
  Interventions: Device: Ablation

INTERVENTIONS:
Device: Ablation — Ablation of a single-side of the greater splanchnic nerve

SUMMARY:
The purpose of this study is to evaluate the safety and potential benefits of single-side block of a nerve that connects to the intestines, liver and spleen called the "greater splanchnic nerve" for the treatments of patients with symptomatic heart failure who have normal pumping of the heart. The study will be performed in patients whose heart failure is not responding well to standard treatments and remain symptomatic.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic heart failure
* Transthoracic echocardiographic evidence of diastolic dysfunction
* Ongoing stable GDMT HF management and management of potential comorbidities
* LVEF ≥50% in the past 3 months

Key Exclusion Criteria:

* Cardiac resynchronization therapy initiated within the past 6 months
* Advanced heart failure
* Admission for HF within the past 30 days
* Presence of significant valve disease
* Mean right atrial pressure (RAP) >20mmHg during hemodynamic screening

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Composite incidence of one or more of the following: major adverse cardiac, cerebrovascular embolic, or renal event (MACCRE) | 1 month
  Composite incidence of one or more of the following: major adverse cardiac, cerebrovascular embolic, or renal event (MACCRE) through 1-month follow up based on Independent Physician Adjudicator (IPA) assessment:
  Cardiovascular death; Embolic stroke; Device or procedure-related adverse cardiac events
Mean change of PCWP with exercise after index procedure ablation as compared to baseline | 1 month
  Mean change of PCWP with exercise after index procedure ablation as compared to baseline

SECONDARY OUTCOMES:
Incidence of MACCRE, all serious adverse events, all-cause mortality, CV mortality and HF related mortality | 6 month
  Incidence of MACCRE, all serious adverse events, all-cause mortality, CV mortality and HF related mortality
Change in average PCWP as compared to baseline | 1 month
  Change in average PCWP as compared to baseline
Secondary Efficacy Endpoint | 1, 3, 6 months
  Change in the quality of life according to the Kansas City Cardiomyopathy Questionnaire (KCCQ) between baseline and follow-up
Secondary Efficacy Endpoint | 1, 3, 6 months
  Change in exercise tolerance as measured by the 6 minute walk test (6MWT) between baseline and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Howard Levin, MD, Study Chair — Coridea, Inc.
Locations (3):
- Nemocnice Na Homolce, Prague, Czechia
- Georgia (2):
  - Tbilisi Heart and Vascular Clinic, Tbilisi
  - Tbilisi Heart Center, Tbilisi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fudim M, Zirakashvili T, Shaburishvili N, Shaishmelashvili G, Sievert H, Sievert K, Reddy VY, Engelman ZJ, Burkhoff D, Shaburishvili T, Shah SJ. Transvenous Right Greater Splanchnic Nerve Ablation in Heart Failure and Preserved Ejection Fraction: First-in-Human Study. JACC Heart Fail. 2022 Oct;10(10):744-752. doi: 10.1016/j.jchf.2022.05.009. Epub 2022 Jul 6. PMID 36175060